CLINICAL TRIAL: NCT04565990
Title: A Multicenter, Single-arm, Open-label, Long-term Follow-up Safety Study of Selexipag in Participants Who Participated in a Previous Selexipag Study
Brief Title: A Study of Selexipag in Participants Who Participated in a Previous Selexipag Study
Acronym: SOMBRERO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108892; 2020-000475-21 (EudraCT Number); 67896049PUH3001 (Other: Actelion)
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selexipag (Experimental): Participants will receive selexipag tablets twice daily with the dose strength corresponding to their individual maximum tolerated dose (iMTD) from the parent study.
  Interventions: Drug: Selexipag

INTERVENTIONS:
Drug: Selexipag — Selexipag tablets will be administered orally at all dose strengths (200, 400, 600, 800, 1000, 1200, 1400 and 1600 microgram) twice daily.
  Other Names: JNJ-67896049; ACT-293987

SUMMARY:
The purpose of this study is to assess the long-term safety of selexipag while providing continued selexipag treatment for participants who were previously enrolled in an Actelion-sponsored study with selexipag and who derived benefit from selexipag in indications for which a positive benefit-risk has been established.

ELIGIBILITY:
Inclusion Criteria:

* Treated with selexipag at the end of a parent study and: a) the parent study has established efficacy with a favorable benefit/risk profile for the indication under investigation; b) participant may continue to benefit from treatment with selexipag; c) has completed the end of treatment (EOT) visit of the parent study; d) no alternative means of access to selexipag have been identified
* Women of childbearing potential must use an acceptable method of contraception throughout the study and until at least 1 month following the last dose of study intervention
* Women of childbearing potential must have a negative urine (or serum if applicable) pregnancy test at screening on Day 1 or at the last visit of the parent study
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Suspected or known pulmonary veno-occlusive disease
* Known allergies, hypersensitivity, or intolerance to selexipag or its excipients
* Interruption of study intervention for more than 14 days since the last dose of study intervention taken in the parent study
* Female participant being pregnant, or breastfeeding, or planning to become pregnant at the time of screening and while enrolled in this study
* Uncontrolled thyroid disease
* Known and documented severe hepatic impairment, example, Child-Pugh Class C
* Taken any disallowed therapies, Concomitant Therapy before the planned first dose of study intervention: a) treatment with a strong CYP 2C8 inhibitor (example, gemfibrozil); b) treatment with oral prostacyclin analogs (example, beraprost, treprostinil) since the last dose of study intervention taken in the parent study; c) any investigational treatment other than selexipag
* Severe coronary heart disease or unstable angina, myocardial infarction within the last 6 months, decompensated cardiac failure if not under close medical supervision, severe arrhythmia, cerebrovascular events (example, transient ischemic attack, stroke) within the last 3 months, or congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to PH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (13):
- Belarus (2):
  - The Republican Scientific-Practical Center ''Cardiology'', Minsk
  - Minsk Regional Clinical Hospital, Minsk
- India (2):
  - Sanjivani Hospitals, Ahmedabad
  - Apollo Hospitals, Chennai
- Institutul de pneumoftiziologie Marius Nasta, Bucharest, Romania
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Taiwan (2):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Ukraine (3):
  - Municipal Inst. Of Dnipropetrovsk Region. Council, Dnipro
  - Health Care Municipal Institution City Clinical Hospital #13, Kharkiv
  - State Institute Of Phthisiology And Pulmonology N.A. F.G. Yanovskiy Of Ams Ukraine, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Selexipag: Participants with pulmonary arterial hypertension (PAH) who completed the parent study AC-065A302 (NCT01106014) continued treatment with selexipag in this study (200 to 1600 micrograms [mcg] selexipag tablet orally twice daily [bid]) from Day 1 up to 28 months with the same individual maximum tolerated dose (iMTD) that they were taking at the end of their parent study. Eligible participants were then followed up for safety up to 30 days after the last dose of selexipag.
Period: Overall Study
Arm/Group | Selexipag
Started | 43
Completed | 36
Not Completed | 7
Not completed — Death | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Selexipag
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (13.25)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 37
  From 65 to 84 years | 6
  >=85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  BELARUS | 21
  INDIA | 4
  ROMANIA | 2
  SOUTH KOREA | 4
  TAIWAN | 3
  UKRAINE | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. Adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were defined as AEs occurring at or after the initial administration of study intervention through the day of last dose plus 3 days. Data includes all TEAEs irrespective of whether they were serious or non-serious.
Time Frame: From Day 1 up to 3 days after last dose of drug (up to 28 months 3 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention in this study..
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 43
Participants | 22

2. Primary Outcome: Number of Participants With TEAEs Leading to Premature Discontinuation of Selexipag
Description: Number of participants with TEAEs leading to premature discontinuation of selexipag were reported. AE was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were defined as AEs occurring at or after the initial administration of study intervention through the day of last dose plus 3 days.
Time Frame: From Day 1 up to 3 days after last dose of drug (up to 28 months 3 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 43
Participants | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: Number of participants with TESAEs were reported. AE was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. A SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or resulted in congenital anomaly/birth defect. TESAEs were defined as TSAEs occurring at or after the initial administration of study intervention through the day of last dose plus 3 days.
Time Frame: From Day 1 up to 3 days after last dose of drug (up to 28 months 3 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 43
Participants | 7

4. Primary Outcome: Number of Participants With Treatment-emergent Deaths
Description: Number of participants with treatment-emergent deaths during the study were reported.
Time Frame: From Day 1 up to 3 days after last dose of drug (up to 28 months 3 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 43
Participants | 5

5. Primary Outcome: Number of Pregnant Females With Maternal Exposure to Selexipag
Description: Number of pregnant females with maternal exposure to selexipag were reported.
Time Frame: From Day 1 up to 30 days after last dose of drug (up to 29 months)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention in this study. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 36
Participants | 0

ADVERSE EVENTS:
Time Frame: All cause mortality: From Day 1 up to 30 days after last dose of drug (up to 29 months), Other AEs and SAEs: From Day 1 up to 3 days after last dose of drug (up to 28 months 3 days)
Description: Safety analysis set included all enrolled participants who received at least 1 dose of study intervention in this study.
Arm/Group | Selexipag
All-Cause Mortality (participants affected / at risk) | 5/43
Serious Adverse Events (participants affected / at risk) | 7/43
Other Adverse Events (participants affected / at risk) | 20/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selexipag (N=43)
Cardiac Failure Acute (Cardiac disorders) | 1
Covid-19 Pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Subacute Endocarditis (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 1
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selexipag (N=43)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Chronic Gastritis (Gastrointestinal disorders) | 2
Gastric Mucosa Erythema (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Autoimmune Hepatitis (Hepatobiliary disorders) | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 1
Non-Alcoholic Fatty Liver (Hepatobiliary disorders) | 1
Steatohepatitis (Hepatobiliary disorders) | 1
Influenza (Infections and infestations) | 1
Otitis Media Acute (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 4
Rib Fracture (Injury, poisoning and procedural complications) | 1
Vaccination Complication (Injury, poisoning and procedural complications) | 1
Complement Factor C3 Decreased (Investigations) | 1
Complement Factor C4 Decreased (Investigations) | 1
Double Stranded Dna Antibody Positive (Investigations) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Benign Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04565990/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT04565990/SAP_001.pdf